CLINICAL TRIAL: NCT06668948
Title: The Prognostic Role of Fibrinogen to Albumin Ratio in Acute Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelraouf Aboeladab Elnaggar, dr asmaa abdelraouf, Assiut University
Other Study IDs: fibrinogen to albumin ratio
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Patients with Acute Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with acute leukemia

SUMMARY:
The study aim to investigate whether levels of acute phase reactants at diagnosis and after 6 months of follow-up correlate with survival and response to treatment in newly diagnosed acute leukemia.Ultimately, we will evaluate the fibrinogen/albumin ratio, a simple score based on acute phase protein levels, whether it can provide relevant prognostic information in acute leukemia patients at diagnosis and after 6 months of follow-up.

DETAILED DESCRIPTION:
Leukemia is a heterogeneous group of hematologic malignancies that arise from the dysfunctional proliferation of developing leukocytes. It is classified as either acute or chronic based on the rapidity of proliferation and as myelocytic or lymphocytic based on the cell of origin.(Chennamadhavuni et al., 2024) .

Acute myeloid leukemia (AML) is a disease of the bone marrow, a disorder of hematopoietic stem cells due to genetic alterations in blood cell precursors resulting in overproduction of neoplastic clonal myeloid stem cells.(Grimwade D HB, Ivey A. Molecular landscape of acute myeloid leukemia in younger adults and its clinical relevance. Blood. 2016;127).It is the most common acute leukemia in adults and it is the most aggressive cancer with a variable prognosis depending upon the molecular subtypes.(Arber et al., 2016) Acute lymphoblastic leukemia (ALL) is the most common leukemia in the pediatric population, accounting for up to 80% of cases in this group vs. 20% of cases in adults. (Arber et al., 2016). It is a malignancy of B or T lymphoblasts characterized by uncontrolled proliferation of abnormal, immature lymphocytes and their progenitors.(Puckett and Chan, 2024).

Clinical presentation can be nonspecific and span a spectrum of symptoms and signs. The majority of patients present with fever, pallor, and bruising as early signs of marrow suppression or hematologic abnormalities, whereas over 60% can demonstrate organomegaly (spleen and liver). A significant number will have a history of recurrent infections, fatigue, lymphadenopathy, and skin rashes (Clarke RT, Van den Bruel A, Bankhead. 2016)

The complicated interplay between inflammation and cancer development was first proposed in the nineteenth century(Coussens and Werb 2002).Also chronic inflammation promotes carcinogenesis, chemoresistance as well as regional or distal metastasis(Zitvogel, Pietrocola et al. 2017).Furthermore, Malnutrition damages the anatomic barriers, immunity and other defense mechanisms(Ataseven, du Bois et al. 2015).

As a result, the involvement of acute phase proteins has been studied not just during inflammatory illnesses, but also in cancers. Fibrinogen is an acute phase reactant produced by hepatocytes in response to tissue damage or infection via interleukin (IL) (namely IL-6 and IL-1) and tumor necrosis factor-alpha signaling pathways(Gabay and Kushner 1999).

These mediators are upregulated during inflammatory processes, while "negative" acute phase reactants, like transferrin and serum albumin, are downregulated because of decreased synthesis or increased breakdown(Pepys and Hirschfield 2003).

Fibrinogen is a crucial component of the coagulation cascade because it promotes platelet aggregation and acts as a substrate for the production of clots when thrombin converts it to fibrin(Weisel, Phillips Jr et al. 1983).

Plasma fibrinogen levels have been linked to tumor growth and prognosis in several malignancies, including colorectal, endometrial, hepatocellular, and pancreatic (Gan, Yi et al. 2018). The liver produces albumin, which is considered a negative acute phase protein(Spinella, Sawhney et al. 2016).

Plasma albumin regulates plasma osmotic pressure, antioxidant levels, capillary permeability, and immunological function(Arabi, Asiri et al. 2020).

An increasing number of studies have found a link between plasma albumin levels, inflammation, and cancer(Dupré and Malik 2018).

Hypoproteinemia is highly related with poor quality of life in cancer patients and poor prognosis in individuals with a variety of malignancies (Murakawa, Yamamoto et al. 2020).

High fibrinogen and low albumin levels are connected with a bad prognosis in cancer patients(Sohda, Sakai et al. 2022).

The fibrinogen-to-albumin ratio (FAR), a new independent predictor that is both simple and effective, has a higher predictive value than either low serum albumin or high fibrinogen. FAR has been identified as a possible predictor of unfavorable outcomes in a number of cancers(Tan, Zhang et al. 2017).

It was found that high fibrinogen levels were related with poor survival innewly diagnosed leukemia patients (Berger, Heini et al. 2017).

The fibrinogen/albumin ratio (FAR) has emerged as a valuable biomarker reflecting both inflammatory and nutritional status, both of which are critical factors in cancer prognosis. In all types of acute leukemia, the interplay between systemic inflammation and compromised nutritional health is particularly pronounced due to the nature of the disease and the intensity of treatments. Elevated fibrinogen, a key acute phase reactant, is associated with tumor progression, increased coagulation, and worse survival outcomes in malignancies, including leukemia. Meanwhile, albumin serves as a negative acute phase protein, with low levels indicating poor nutritional status and higher inflammatory burdens. The combination of these two markers in the form of the FAR provides a more comprehensive measure of a patient's health than either marker alone(Zhang and Xiao 2019).

FAR consists of fibrinogen and albumin, both of which are commonly used laboratory tests that are easy and inexpensive to obtain. In the future, if FAR can be used in clinical treatment, it will improve the efficiency of diagnosis and reduce the cost of treatment for cancer patients.(Li et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Newly diagnosed patients with acuteleukemia
  2. Not received any treatment

Exclusion Criteria:

* Exclusion criteria:

  1. Patients with chronic inflammatory diseases (e.g., rheumatoid arthritisinflammatory bowel disease) or acute infections that may affect acute phase protein levels.
  2. Patients under chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Newly diagnosed patients with acuteleukemia
  2. Not received any treatment
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The prognostic role of fibrinogen to albumin ratio in acute leukemia patients | 2025

IPD SHARING:
Plan to Share IPD: No